CLINICAL TRIAL: NCT05829720
Title: A Double-blind, Parallel Designed, Randomized Controlled Trial to Investigate Effects of Conventional Vs A2 Milk on Breastmilk Composition and Subsequent Infant Gut Health, Crying and Sleep Patterns in Healthy, Full-term Infants
Brief Title: Investigate Effects of A2 Milk on Breastmilk Composition and Subsequent Infant Gut Health, Crying and Sleep Patterns in Healthy, Full-term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-SM-12-A2-001
Record Dates: First submitted 2023-04-03; First posted 2023-04-26 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Digestive System Disease; Sleepiness; Crying
Keywords: A2 Full Cream Milk; Breastmilk Composition; Gut Health
MeSH Terms: conditions — Digestive System Diseases; Sleepiness; Crying

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- a2 Full Cream Milk (Active Comparator): a2 Full Cream Milk, 200ml/bag, per 100ml serving Nutrient Composition Energy: 250 kcal Protein:3.2g Fat:3.3g Carbohydrate:4.3g Sodium:40mg Calcium:104mg
  Interventions: Dietary Supplement: a2 Full Cream Milk
- Conventional Milk (Weidendorf) (Active Comparator): Conventional Milk (Weidendorf), 200ml/bag,per 100ml serving Nutrient Composition Energy: 267 kcal Protein:3.3g Fat:3.5g Carbohydrate:4.8g Sodium:50mg Calcium:120mg
  Interventions: Dietary Supplement: Conventional Milk (Weidendorf)

INTERVENTIONS:
Dietary Supplement: a2 Full Cream Milk — Mothers in this arm will drink a2 Full Cream Milk twice a day, 200ml each time, for 14 consecutive days. Infants in this arm will be fed with mather's breastmilk exclusively.
  Arms: a2 Full Cream Milk
Dietary Supplement: Conventional Milk (Weidendorf) — Mothers in this arm will drink Conventional Milk (Weidendorf) twice a day, 200ml each time, for 14 consecutive days. Infants in this arm will be fed with mather's breastmilk exclusively.
  Arms: Conventional Milk (Weidendorf)

SUMMARY:
The goal of this interventional study is to investigate effects of a2 Full Cream Milk on Breastmilk composition and subsequent Infant gut health, crying frequency and sleep patterns in Healthy Full-term Infants.

50 mothers and thier infants will be enrolled into 2 study sites, mother and her child as one subject will be randomized to 2 groups for assigned interventions, a2 Full Cream Milk and conventional Milk (Weidendorf). The study will continue for 14 days, and 3 site visits will be made duing the study period. All data specified in the protocol will be captured and recorded into CTMS for analysis.

Researchers will compare the two groups of participants to see if a2 Full Cream Milk has significantly better breastmilk composition and improve infant's gut health, crying frequency and sleep patterns.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who are 25 to 45 years old;
* Mothers who are exclusively breastfeeding with healthy and full-term infants;
* Infants of these mothers who have been exclusively breastfed since birth, and their parent(s) decides to continue exclusively breastfeeding until at least 120 days of age, birth weight between 2500g and 4500g;
* Willing to sign ICF before the study launched.

Exclusion Criteria:

* Mothers with infection or have recently taken the flu / covid vaccine in the last 4 weeks;
* Infant with inborn malformation and with hereditary and/or chronic and/or inborn diseases that could interfere with the survey;
* Evidence of feeding difficulties or intolerance/allergy to cow's milk (mixed-fed group only);
* Conditions requiring infant feedings other than those specified in the protocol;
* Significant systemic disorders (cardiac, respiratory, endocrinological, hematologic, gastrointestinal, or other); or parental refusal to participate;
* Infants with an acute infection or gastroenteritis at time of enrollment;
* Participation in another clinical trial;
* Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Mothers who are exclusively breastfeeding with healthy and full-term infants, infants as participants can be male or female.
Enrollment: 100 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Breast milk excretion of Human Milk oligosaccharide content (HMO) content | Baseline (T0)
  Qualitative analysis of Breast milk excretion of Human Milk oligosaccharide content (HMO) content on baseline day
Breast milk excretion of Human Milk oligosaccharide content (HMO) content | After 14 days of supplementation (T14)
  Qualitative analysis of Breast milk excretion of Human Milk oligosaccharide content (HMO) content on day 14
Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score | Baseline (T0)
  Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score, range 10 to 60
Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score | After 14 days of supplementation (T14)
  Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score, range 10 to 60

SECONDARY OUTCOMES:
Infant Crying Frequency | baseline day, to day 14
  The Frequency of Infant Crying Daily
Number of Hours of Infants Sleeping | baseline day, to day 14
  Number of Hours of Infants Sleeping Daily

CONTACTS AND LOCATIONS:
Overall Officials: Zhixu Wang, MD, Principal Investigator — School of Public Health, Nanjing Medical University; Fan Yang, PhD, Principal Investigator — West China Second Hospital, Sichuan University; Yi Sun, MD, Principal Investigator — Shanghai Tongren Hospital
Locations (2):
- China (2):
  - Jinhua Wenrong Hospital, Jinhua, Zhejiang
  - Qiu Bin Community Hospital, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jianqin S, Leiming X, Lu X, Yelland GW, Ni J, Clarke AJ. Effects of milk containing only A2 beta casein versus milk containing both A1 and A2 beta casein proteins on gastrointestinal physiology, symptoms of discomfort, and cognitive behavior of people with self-reported intolerance to traditional cows' milk. Nutr J. 2016 Apr 2;15:35. doi: 10.1186/s12937-016-0147-z. PMID 27039383
- [Background] He M, Sun J, Jiang ZQ, Yang YX. Effects of cow's milk beta-casein variants on symptoms of milk intolerance in Chinese adults: a multicentre, randomised controlled study. Nutr J. 2017 Oct 25;16(1):72. doi: 10.1186/s12937-017-0275-0. PMID 29070042
- [Background] Sheng X, Li Z, Ni J, Yelland G. Effects of Conventional Milk Versus Milk Containing Only A2 beta-Casein on Digestion in Chinese Children: A Randomized Study. J Pediatr Gastroenterol Nutr. 2019 Sep;69(3):375-382. doi: 10.1097/MPG.0000000000002437. PMID 31305326
- [Background] Sheng XY, Buthmanaban V, van Lieshout GAA, Parikh P. Reduced Occurrence of Gastrointestinal Symptoms in Chinese Infants Fed Minimally Processed Commercially Available Formula: A Cross-Sectional Observational Study. J Nutr Metab. 2020 Mar 25;2020:1807397. doi: 10.1155/2020/1807397. eCollection 2020. PMID 32300486
- [Background] Iacono G, Merolla R, D'Amico D, Bonci E, Cavataio F, Di Prima L, Scalici C, Indinnimeo L, Averna MR, Carroccio A; Paediatric Study Group on Gastrointestinal Symptoms in Infancy. Gastrointestinal symptoms in infancy: a population-based prospective study. Dig Liver Dis. 2005 Jun;37(6):432-8. doi: 10.1016/j.dld.2005.01.009. Epub 2005 Mar 2. PMID 15893282
- [Background] van de Heijning BJ, Berton A, Bouritius H, Goulet O. GI symptoms in infants are a potential target for fermented infant milk formulae: a review. Nutrients. 2014 Sep 25;6(9):3942-67. doi: 10.3390/nu6093942. PMID 25255831
- [Background] Ferreira-Maia AP, Matijasevich A, Wang YP. Epidemiology of functional gastrointestinal disorders in infants and toddlers: A systematic review. World J Gastroenterol. 2016 Jul 28;22(28):6547-58. doi: 10.3748/wjg.v22.i28.6547. PMID 27605889
- [Background] Vandenplas Y, Abkari A, Bellaiche M, Benninga M, Chouraqui JP, Cokura F, Harb T, Hegar B, Lifschitz C, Ludwig T, Miqdady M, de Morais MB, Osatakul S, Salvatore S, Shamir R, Staiano A, Szajewska H, Thapar N. Prevalence and Health Outcomes of Functional Gastrointestinal Symptoms in Infants From Birth to 12 Months of Age. J Pediatr Gastroenterol Nutr. 2015 Nov;61(5):531-7. doi: 10.1097/MPG.0000000000000949. PMID 26308317
- [Background] Shamir R, St James-Roberts I, Di Lorenzo C, Burns AJ, Thapar N, Indrio F, Riezzo G, Raimondi F, Di Mauro A, Francavilla R, Leuchter RH, Darque A, Huppi PS, Heine RG, Bellaiche M, Levy M, Jung C, Alvarez M, Hovish K. Infant crying, colic, and gastrointestinal discomfort in early childhood: a review of the evidence and most plausible mechanisms. J Pediatr Gastroenterol Nutr. 2013 Dec;57 Suppl 1:S1-45. doi: 10.1097/MPG.0b013e3182a154ff. No abstract available. PMID 24356023
- [Background] Ul Haq MR, Kapila R, Sharma R, Saliganti V, Kapila S. Comparative evaluation of cow beta-casein variants (A1/A2) consumption on Th2-mediated inflammatory response in mouse gut. Eur J Nutr. 2014 Jun;53(4):1039-49. doi: 10.1007/s00394-013-0606-7. Epub 2013 Oct 29. PMID 24166511